CLINICAL TRIAL: NCT04854070
Title: Intravascular Ultrasound Guidance for Complex High-risk Indicated Procedures
Acronym: IVUS-CHIP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ECRI bv (Industry)
Collaborators: Boston Scientific Corporation (Industry); Cardialysis B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ECRI-14
Record Dates: First submitted 2021-04-08; First posted 2021-04-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Complex Coronary Lesions
Keywords: Percutaneous coronary intervention; Angiographic guided PCI; Intra-vascular ultrasound guided PCI

STUDY DESIGN:
Intervention Model Description: Randomization in a 1:1 fashion to IVUS-guided PCI versus angio-guided PCI
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- IVUS-guided PCI (Experimental): Method is already used in standard care, but in this trial compared to another method also already used in standard care
  Interventions: Device: IVUS
- Angio-guided PCI (Active Comparator): Method is standard care
  Interventions: Device: Angio

INTERVENTIONS:
Device: IVUS — IVUS-guided approach in patients with complex coronary lesions undergoing PCI
  Arms: IVUS-guided PCI
Device: Angio — Angio-guided approach in patients with complex coronary lesions undergoing PCI
  Arms: Angio-guided PCI

SUMMARY:
The IVUS CHIP trial is a post-marketing strategy study in which patients with complex coronary lesions, undergoing percutaneous coronary intervention (PCI), are treated either with intravascular ultrasound (IVUS) guided PCI or angiographic guided PCI .

The IVUS-guided PCI approach is indicated to reduce the frequency of target-lesion failure (cardiac death, target-vessel myocardial infarction, and clinically indicated target-lesion revascularization) in patients with complex coronary lesions undergoing PCI.

The objective of this study is to assess the superiority of an IVUS-guided approach versus an angio-guided approach in patients with complex coronary lesions undergoing PCI.

DETAILED DESCRIPTION:
During percutaneous coronary intervention (PCI) coronary arteries are visualized to guide placing the stent. In this study 2 currently utilized methods of visualizing coronary arteries during PCI are compared: intravascular ultrasound (IVUS) and angiographic guided PCI for patients with complex coronary lesions. The use of IVUS during PCI is suggested to give better results than angiographic guided PCI.

The IVUS-CHIP trial is a randomized, controlled, multicenter, international, post-marketing study. A total of 2020 patients, in 7 European countries and approximately 40 hospitals, will be included, randomized in a 1:1 fashion to IVUS-guided PCI versus angio-guided PCI, and followed up for at least 2 years.

The IVUS-CHIP is an event-driven study; primary analysis of the data will take place after at least 169 patients have experienced an event.

ELIGIBILITY:
Inclusion Criteria:

All of the following:

1. The patient must be ≥18 years of age
2. Patients with an indication for PCI of at least one lesion satisfying any of the following criteria:

   1. Angiographic heavy calcification
   2. Ostial lesions
   3. True bifurcation lesions involving side-branches >2.5mm
   4. Left main lesions
   5. Chronic total occlusion
   6. In-stent restenosis
   7. Long-lesions (estimated stent length > 28mm) OR Patient with an indication for PCI for any lesion and in need for elective mechanical circulatory support assisted PCI
3. Presenting with silent ischemia, stable angina, unstable angina or non-ST-elevation acute coronary syndrome (NSTE-ACS)
4. All lesions must be suitable for treatment with the Synergy stent system, Synergy Megatron system, or other Synergy platform iteration
5. The patient is willing and able to cooperate with study procedures and follow-up until study completion
6. Subject is able to confirm understanding of risks, benefits and treatment alternatives and he/she provides informed consent prior to any protocol-related procedure, as approved by the appropriate Ethics Committee

Exclusion Criteria:

Any of the following:

1. ST-elevation myocardial infarction, cardiogenic shock
2. Known untreated severe valvular heart disease
3. IVUS is strictly required for pre-PCI lesion severity assessment
4. Known contraindication or hypersensitivity to everolimus, platinum-chromium, or to anticoagulants
5. Absolute contraindications or allergy that cannot be pre-medicated, to iodinated contrast or to antiplatelet drugs, including both aspirin and P2Y12 inhibitors
6. Non-cardiac co-morbidities with a life expectancy less than 1 year
7. Currently participating in another trial that is not yet at its primary endpoint. The patient is not allowed to participate in another investigational device or drug study until the trial primary endpoint time point is achieved and may only be enrolled once in the study
8. Women of childbearing potential who do not have a negative pregnancy test within 7 days before the procedure and women who are breastfeeding
9. Subject belongs to a vulnerable population (per investigator's judgment) or subject unable to read or write

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2020 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Target-vessel failure comparison of IVUS-guided PCI to angio-guided PCI in patients with complex coronary lesions | From date of randomization until the analysis cut-off date at approximately 15-18 months of median follow-up
  Target-vessel failure is defined as a composite of cardiac death, target vessel myocardial infarction, or clinically indicated target-vessel revascularization

SECONDARY OUTCOMES:
Composite of target-vessel myocardial infarction and clinically indicated target vessel revascularization | From date of randomization until the analysis cut-off date at approximately 15-18 months of median follow-up
  Composite of target-vessel myocardial infarction and clinically indicated target vessel revascularization
Clinically-indicated target vessel revascularization | From date of randomization until the analysis cut-off date at approximately 15-18 months of median follow-up
  Clinically-indiated target vessel revascularization is defined as any clinically-indicated repeat percutaneous intervention or surgical bypass of any segment of the target vessel
Composite of cardiac death and target-vessel myocardial infarction | From date of randomization until the analysis cut-off date at approximately 15-18 months of median follow-up
  Composite of cardiac death and target-vessel myocardial infarction
Target-Lesion Failure (TLF) | From date of randomization until the analysis cut-off date at approximately 15-18 months of median follow-up
  Target-Lesion Failure is defined as a composite of cardiac death, target vessel myocardial infarction, or clinically indicated target-lesion revascularization
Target-lesion revascularization | From date of randomization until the analysis cut-off date at approximately 15-18 months of median follow-up
  Target-lesion revascularization is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion
Cardiac death | From date of randomization until the analysis cut-off date at approximately 15-18 months of median follow-up
  Cardiac death is defined as death resulting from cardiovascular causes

CONTACTS AND LOCATIONS:
Overall Officials: R. Diletti, Dr., Principal Investigator — Erasmus Medical Center
Locations (37):
- Belgium (4):
  - OLVZ, Aalst
  - CHU, Charleroi
  - ZOL Sint-Jan, Genk
  - University Hospital Gasthuisberg, Leuven
- France (7):
  - Clinique Saint-Augustin, Bordeaux
  - Cardiovascular Institute of Grenoble, GHM, Grenoble
  - Hopital Privé Jacques Cartier, Massy
  - Centre Cardiologique du Nord Saint-Denis, Saint-Denis
  - CHU, Toulouse
  - Clinique Pasteur, Toulouse
  - CHRU Tours - HopitalTrousseau, Tours
- Germany (6):
  - Segeberger Kliniken, Bad Segeberg
  - Charite Universitatsmedizin Berlin, Berlin
  - Heart Center Dresden, Dresden
  - Universitätsklinikum Frankfurt, Frankfurt
  - University of Giessen, Giessen
  - MediClin Heartcenter Lahr, Lahr
- Italy (4):
  - University of Ferrara, Ferrara
  - Humanitas Research Hospital, Milan
  - Ospedale degli infermi di Rivoli, Rivoli
  - Ospedale dell'Angelo, Venezia
- Netherlands (5):
  - Noordwest Hospital Group, Alkmaar
  - VuMC, Amsterdam
  - Albert Schweitzer hospital, Dordrecht
  - Catharina hospital, Eindhoven
  - Erasmus University Medical Center, Rotterdam
- Spain (7):
  - Bellvitge University Hospital, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Reina Sofia Hospital, Córdoba
  - Hospital la Paz, Madrid
  - La Princesa University Hospital, Madrid
  - Marques de Valdecilla University Hospital, Santander
  - University Clinical Hospital of Valladolid, Valladolid
- United Kingdom (4):
  - Royal Victoria Hospital, Belfast
  - Golden Jubilee National Hospital, Glasgow
  - St. George's University Hospital, London
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Diletti R, Daemen J, Faurie B, Barbierato M, Tchetche D, Hovasse T, Teeuwen K, Oemrawsingh RM, Allali A, Campo G, Bennett J, Alfonso F, Mashayekhi K, Moreno R, Abdelwahed YS, Dedic A, de la Torre Hernandez JM, Murphy JC, Amat-Santos I, Dens J, Franze A, Leistner D, Ghattas A, Spratt JC, Banning AP, Tijssen JGP, Spitzer E, Van Mieghem NM; IVUS CHIP investigators. Intravascular ultrasound guidance for complex high-risk indicated procedures: The IVUS CHIP trial study design. Am Heart J. 2026 Jan 3;294:107339. doi: 10.1016/j.ahj.2026.107339. Online ahead of print. PMID 41490527